CLINICAL TRIAL: NCT06411106
Title: An Exploratory, Single-center, Two-part Study to Characterize Cutaneous Lupus Erythematosus and Investigate the Effect of an Immune Challenge by Comparing CLE Patients With Healthy Volunteers
Brief Title: Deep Phenotyping of Cutaneous Lupus Erythematosus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHDR2307; NL84645.056.23 (Other: CCMO)
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: CLE; Cutaneous lupus erythematosus; Deep phenotyping; Immune challenge; Healthy volunteers
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Imiquimod

STUDY DESIGN:
Intervention Model Description: Part A of the study is observational and Part B has an intervention. In Part B, the intervention is a challenge with imiquimod. All patients and healthy volunteers will receive the same challenge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Experimental): CDLE patients and healthy volunteers In part B of this study, 5 mg imiquimod (100 mg Aldara®) per skin area (in total two skin areas) will be applied for two consecutive days under occlusion.
  Interventions: Drug: IMIQUIMOD cream 50mg/g

INTERVENTIONS:
Drug: IMIQUIMOD cream 50mg/g — 5 mg imiquimod (100mg Aldara®) per treatment site with a 12mm Finn chamber
  Other Names: Aldara

SUMMARY:
Cutaneous lupus erythematosus (CLE) is an autoimmune disease of which the pathogenesis and pathophysiology are not fully understood. Given the complex and heterogeneous character of the disease, identification, and development of specific biomarkers for diagnosis, disease subtyping, disease severity, and treatment response in CLE is challenging. Therefore, the main objective of the current study is to further characterize CLE by using a deep phenotyping approach. Moreover, the role of TLR7 activation in the pathophysiology of the various clinical subtypes of CLE will be specifically studied. With this approach the investigators aim to characterize objectively measured disease characteristics and detect novel biomarkers for CLE(-subtypes).

DETAILED DESCRIPTION:
Cutaneous lupus erythematosus (CLE) is a rare but burdensome autoimmune disease that includes various subtypes including acute cutaneous LE (ACLE), subacute cutaneous LE (SCLE), intermittent cutaneous LE (ICLE) i.e., lupus tumidus (LET) and chronic cutaneous LE (CCLE). These subtypes differ in lesion morphology and histopathology, however disease stratification is often a challenge.

Knowledge on mechanisms involved in the pathogenesis and pathophysiology of CLE is growing, however much remains unknown. The current concept regarding the onset of the disease comprises a genetic background predisposing to CLE triggered by factors such as UV light, what leads to cellular stress and eventually to the release of DNA components in keratinocytes (Fetter et al., 2022). Activation of both Toll-like receptor (TLR)-dependent and TLR-independent inflammatory signalling cascades leads to increased expression of several cytokines, in particular type I interferon (IFN). Type I interferon mediates increased expression of proinflammatory chemokines via the JAK-STAT pathway, leading to recruitment of immune cells, release of cytokines and a chronic reactivation of innate immune pathways.

Findings on the pathogenesis of the disease have led to the development of several targeted therapies that are currently being investigated in clinical trials. However, blockage of one important pathway might not suffice for decreasing disease activity given the limited efficacy of selective IFN antibodies in clinical trials (Kalunian et al., 2016), (Khamashta et al., 2016) (Werth et al., 2017).

Only few biomarkers for CLE have been validated and widely incorporated into clinical practice (Zhu et al., 2021). Type I interferon-inducible proteins can be potentially used to assess disease severity of SCLE and CDLE (Braunstein et al., 2013). Furthermore, low complement in CLE patients may be related to poor prognosis and increased risk of developing systemic disease (Vera et al., 2010) (Vera et al., 2010).

Therefore, the objectives of the current study are to evaluate disease-related characteristics in CLE patients and to evaluate the variability between patients using a deep phenotyping approach, and to investigate the immune response of CLE patients following an ex vivo and in vivo imiquimod skin challenge. The study consists of an observational (part A) and interventional (part B) part in CLE patients and healthy volunteers.- With this approach the investigators aim to characterize objectively measured disease characteristics and detect novel biomarkers for CLE(-subtypes).

This study is part of the Next Generation Immuno Dermatology consortium SKINERGY trials.

ELIGIBILITY:
Eligible healthy volunteers must meet all the following inclusion criteria at screening:

1. Signed informed consent prior to any study-mandated procedure.
2. Male or female subjects, 18 to 65 years of age at the time of signing informed consent; in general, stable good health as per judgement of the investigator based upon the results of a medical history, physical examination, vital signs, ECG, and laboratory assessments performed at screening. Repeated laboratory testing may be performed at the discretion of the clinical investigator.
3. Body mass index (BMI) > 18.0 and < 32.0 kg/m2
4. Fitzpatrick skin type I-III (Caucasian).
5. Subjects and their partners of childbearing potential must use effective contraception for the duration of the study.
6. No clinically significant skin disease as judged by the investigator.
7. No history of hypertrophic scarring or keloid.
8. Subject is willing to refrain from application of any topical product (e.g., ointments, cream or washing lotions) on the target lesion(s)skin 24 hours prior to every study visit day.
9. Subject has the ability to communicate well with the investigator in the Dutch language and is willing to comply with the study requirements.

Eligible CLE patients must meet all the following inclusion criteria at screening:

1. Signed informed consent prior to any study-mandated procedure.
2. Male or female CLE patients, 18 to 65 years of age at the time of signing informed consent; in general, stable good health as per judgement of the investigator based upon the results of a medical history, physical examination, vital signs, ECG, and laboratory assessments performed at screening. Repeated laboratory testing may be performed at the discretion of the clinical investigators.
3. Body mass index (BMI) > 18.0 and < 35.0 kg/m2.
4. Only applicable for CDLE patients who will also participate in part B: Fitzpatrick skin type I-III (Caucasian).
5. Subjects and their partners of childbearing potential must use effective contraception for the duration of the study.
6. Patient has the ability to communicate well with the investigator in the Dutch language and is willing to comply with the study requirements.
7. Subject is willing to refrain from application of any topical product (e.g., ointments, cream or washing lotions) on the target lesion(s) 24 hours prior to every study visit day.
8. Participants must have a diagnosis of SCLE, CDLE or LET that fulfils the following:

   * Confirmed CLE diagnosis by clinicopathological correlation.
   * At least one CLE skin lesion of at least 3x3 cm suitable as assessed by the investigator for measurements performed in the study.
   * Location of the lesion(s) selected for biopsy outside the face (possible are e.g., neck, chest, back, limbs, scalp, ear etc.).
   * Receiving one of the following systemic treatments for CLE (stable for a minimum of 8 weeks):

     * None
     * Hydroxychloroquine
   * An overall CLE Disease Area and Severity Index Activity (CLASI-A) Score ≥3 without counting any diffuse alopecia or oral ulcers

Eligible healthy volunteers must meet none of the following exclusion criteria at screening:

1. (History of) immunological abnormality (e.g., immune suppression) that may interfere with study objectives, in the opinion of the investigator.
2. Have any current and/or recurrent clinically significant skin condition, including tattoos.
3. Antibiotic use, operation, or clinically significant intervention by surgeon/dentist within one month before Day 1.
4. Positive hepatitis B surface antigen (HbsAg), hepatitis C antibody (HCV ab), or human immunodeficiency virus antibody (HIV ab) at screening.
5. Participation in an investigational drug study within 3 months prior to screening or more than 4 times a year.
6. Loss or donation of blood over 500mL within three months prior to screening.
7. Subject is willing to refrain from the use of any medication within 28 days prior to Day 1, if the investigator judges it may interfere with the study objectives.
8. History of alcohol abuse or consumption exceeding 5 standard drinks per day on average within 3 months of screening.
9. Positive urine test for drugs or history of abuse at screening. Urine drug test may be repeated at the discretion of the investigator.
10. Pregnant, a positive pregnancy test, intending to become pregnant during the study conduct, or breastfeeding.
11. (A history of) any clinically significant medical condition, factor or abnormality that might interfere with study conduct or interpretation, as judged by the investigator.
12. Previous use of Aldara (imiquimod cream) 3 months prior to the Day 1 visit in part B.
13. Any active or chronic and/or uncontrolled condition that, in the opinion of the investigator, may influence study conduct or interpretation

Eligible CLE patients must meet none of the abovementioned and following exclusion criteria at screening:

1. Presence of a relevant skin infection or disease in the target areas other than the observational disease (CLE), inclusively, but not limited to atopic dermatitis, psoriasis vulgaris and dermatomycosis.
2. Having received treatments for CLE or any other disease within the following intervals prior to Day 1:

   1. <2 weeks for topical treatment, e.g., corticosteroids at target area(s)
   2. <6 weeks for systemic therapy with immunosuppressive agents (other than hydroxychloroquine stable use for a minimum of 8 weeks)
   3. <12 weeks for biologics
   4. <8 weeks procedure or surgery in or close to the target areas
   5. <3 months for chemotherapeutical treatment
3. Presence of severe lupus-associated renal disease.
4. Presence of antiphospholipid syndrome.
5. Active or unstable lupus-associated neuropsychiatric disease.
6. Severe organ SLE manifestation(s) (e.g., active myocarditis) or unstable disease as judged by the investigator.
7. Diagnosis of systemic lupus erythematosus (SLE) according to the EULAR-ACR criteria (2019) or substantial indication for systemic involvement (part B only).
8. Low complement (C3 and/or C4) levels at screening (< ULN) (part B only).
9. Positive ANA and anti-dsDNA and/or anti-SM at screening (part B only).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Skin punch biopsies | Day 15
  Skin punch biopsies (4mm) will be taken from (non-)lesional skin and healthy for histology and RNA-sequencing analysis.
3D Multispectral imaging | Day 1 - 15
  The redness and superficial morphology of (non-)lesional skin sites and healthy skin will be determined using a 3D multispectral imaging system.
Laser Speckle Contrast Imaging (LSCI) | Day 1 - 15
  The cutaneous microcirculation of (non-)lesional skin sites and healthy skin will be monitored over a 40 second timespan with a laser speckle contrast imager.
Line-Field Confocal Optical Coherence Tomography (LC-OCT) | Day 1 - 15
  LC-OCT is a non-invasive optical imaging technique based on a combination of the optical principles of optical coherence tomography and reflectance confocal microscopy with line-field illumination, which can generate cell-resolved images of the skin, in vivo, in vertical section, horizontal section and in three dimensions.
Skin barrier function by Trans-Epidermal Water Loss (TEWL) | Day 1 - 15
  The barrier status by trans epidermal water loss of (non-)lesional skin and healthy skin will be determined using TEWL.
Cutaneous microbiome | Day 15
  The cutaneous microbiome of (non-)lesional skin and healthy skin is collected by swabbing.
Lipidomics of the stratum corneum and OLINK | Day 15
  Tape stripping will be performed on (non-)lesional skin and healthy skin for extraction of lipids for analysis and analysis will be performed using OLINK.
Blister immune cell subsets | Day 15
  Blisters will be induced on the (non-)lesional skin and healthy skin, and the blister fluid will be aspirated. The blister fluid will be analyzed for the presence of immune cells using flow cytometry.
Faecal microbiome (optional for patients) | Day 15
  The bacterial composition of a stool samples will be determined.
Circulating cytokines | Day 15
  Blood will be drawn using a venipuncture and analyzed for cytokines.
Interferon (IFN) signature | Day 15
  Blood will be drawn using a venipuncture and analyzed for gene expression related to interferon (IFN).
User experience and subjective burden questionnaire | Day 15
  Measures the user experience and subjective burden of the different assessments performed in this study.

SECONDARY OUTCOMES:
Ex vivo response to imiquimod | Day 15
  Blood will be collected at one timepoint and stimulated ex vivo with imiquimod for cytokine analysis.
In vivo response to imiquimod | Day 1 - 4 (Part B)
  After topical application of imiquimod for 2 consecutive days, the skin response will be assessed by imaging techniques (multispectral 3D, 2D, LSCI, LC OCT and TEWL) and a skin punch biopsy will be collected 48h after the first application. Blood for circulating cytokine analysis, complement, and autoantibodies will be collected and compared to the baseline sample (taken during part A).
Patient reported outcomes | Day 1- 4 (Part B)
  Patients will be asked to report on their itch and pain using a Numeric Rating Scale (NRS).

CONTACTS AND LOCATIONS:
Overall Officials: R. Rissmann, RPh, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No